CLINICAL TRIAL: NCT06205654
Title: Invloed Van Verlichting (en Daglicht) Op Bewoners Met Dementie in Woonzorgcentra
Brief Title: Effect of Improved Indoor Lighting on Residents of Residential Care Homes with Dementia
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Odisee University College (Unknown)
Responsible Party: Principal Investigator, Wouter Ryckaert, Prof. Dr., KU Leuven
Other Study IDs: S66305
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Dementia
Keywords: Lighting; Integrative lighting; Dementia; Nursing home; Residential care home
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: innovative lighting designs are implemented in the living area.
- Control: no significant modifications to their lighting conditions are implemented in the living area

SUMMARY:
Elderly with dementia living in residential care homes often have limited access to adequate lighting (daylight). Light can however positively impact the individual on a number of factors, including sleep quality and mental health. The proposed non-invasive study seeks to evaluate the impact of an improved lighting environment in the living areas of residential care home residents with dementia on both the physical and mental well-being of these individuals. To assess sleep quality, an actigraphy device will be used from which a number of parameters corresponding to sleep quality can be obtained. Mental health/behaviour of the participants will be assessed by validated questionnaires. These questionnaires will be filled for each participant independently by 2 members of the nursing staff.

Two groups of residential care home residents will be observed during this study: an intervention group and a control group. In the intervention group, innovative lighting designs are already implemented in the living area. The control group will experience no significant modifications to their lighting conditions. Extra luminaires (floor lamp/table lamp) will be employed without significantly improving the light exposure during the day.

It is hypothesized that the introduction of enhanced lighting during the day in the living area of the intervention group will result in improved sleep quality and enhanced mental well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with dementia
2. Residing in the selected living area

Exclusion Criteria:

1. Blind individuals
2. Not residing in the selected living area
3. Not diagnosed with dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two residential care homes are participating in this study. In one residential care home, improved lighting was implemented in two living rooms. The intervention group consists of participants living in one of these living rooms. The control group consists of participants living in the other residential care home (where improved lighting was not implemented).
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in sleep efficiency at Week 15 | Baseline + Week 15
  Sleep efficiency is the actual sleep time expressed as a percentage of time in bed as measured by actigraphy. Higher percentage indicates better sleep efficiency.
  Change = percentage point difference between Baseline and Week 15
Change from Baseline in Fragmentation Index at Week 15 | Baseline + Week 15
  The Fragmentation Index is an indication of the degree of fragmentation of the sleep period, and can be used as an indication of sleep quality. This parameter is measured using actigraphy.
  Change = (Week 15 Fragmentation Index - Baseline Fragmentation Index)
Change from Baseline in interdaily stability at Week 15 | Baseline + Week 15
  Interdaily stability quantifies the degree of regularity in the activity-rest pattern. Range of 0 to 1 where a value of 0 indicates a total lack of rhythm and a value of 1 indicates a perfectly stable rhythm. This parameter is measured using actigraphy.
  Change = (Week 15 Interdaily stability - Baseline Interdaily stability)
Change from Baseline in Intradaily variability at Week 15 | Baseline + Week 15
  Intradaily variability quantifies the degree of fragmentation of activity-rest periods. The variable has a theoretical range of 0 to 2 with higher values indicating higher fragmentation. Typical values for healthy subjects will be below 1. This parameter is measured using actigraphy.
  Change = (Week 15 Intradaily variability - Baseline Intradaily variability)
Change from Baseline in L5 average at Week 15 | Baseline + Week 15
  L5 average provides the average activity level for the sequence of the least five active hours.This value provides an indication of how restful (inactive) and regular the sleep periods are. This parameter is measured using actigraphy.
  Change = (Week 15 L5 average - Baseline L5 average)
Change from Baseline in M10 average at Week 15 | Baseline + Week 15
  M10 average provides the average activity level for the sequence of the highest (most) ten active hours. This value provides an indication of how active and regular the wake periods are. This parameter is measured using actigraphy.
  Change = (Week 15 M10 average - Baseline M10 average)
Change from Baseline in number of naps at Week 15 | Baseline + Week 15
  Average number of naps during the day. More naps during the day indicate poorer sleep patterns. This parameter is measured using actigraphy.
  Change = (Week 15 number of naps - Baseline number of naps)
Change from Baseline in agitation on the Cohen-Mansfield Agitation Inventory at Week 15 | Baseline + Week 15
  The Cohen-Mansfield Agitation Inventory is used to assess agitation. It consists of 29 items regarding the manifestation of physically aggressive, physically non-aggressive and verbally agitated behaviors which are scored on a 7-point scale ranging from "Never" to "Several times per hour". The questionnaire is completed for each participant independently by 2 members of the nursing staff.
  Change = (Week 15 score - Baseline score)
Change from Baseline in depression on the Cornell Scale for Depression in Dementia at Week 15 | Baseline + Week 15
  The Cornell Scale for Depression in Dementia is used to assess symptoms of depression in participants with dementia. It consists of different items where each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 as a rule are associated with absence of significant depressive symptoms.
  The questionnaire is completed for each participant independently by 2 members of the nursing staff.
  Change = (Week 15 score - Baseline score)
Change from Baseline in pain on the Doloplus Scale-2 at Week 15 | Baseline + Week 15
  The Doloplus Scale-2 is used to assess pain and the impact of pain. The items are rated for severity on a scale of 0-3 (0=absent, 3=almost always present).
  The questionnaire is completed for each participant independently by 2 members of the nursing staff.
  Change = (Week 15 score - Baseline score)
Change from Baseline in neuropsychiatric symptoms on the Neuropsychiatric Inventory at Week 15 | Baseline + Week 15
  The Neuropsychiatric Inventory (NPI) is used to assess a broad spectrum of neuropsychiatric symptoms, including hallucinations, delusions, and anxiety. The NPI examines 12 sub-domains of behavioral functioning: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances, and appetite and eating abnormalities The questionnaire is completed for each participant independently by 2 members of the nursing staff.
  Change = (Week 15 score - Baseline score)

SECONDARY OUTCOMES:
Age of participant | Baseline measurement
  Age of participant at Baseline
Gender of participant | Baseline measurement
  Gender of participant at Baseline
Length of stay in the nursing home of participant | Baseline measurement
  Length of stay in the nursing home of participant at Baseline
Marital status of participant | Baseline measurement
  Marital status of participant at Baseline
Frequency of visitors of participant | Baseline measurement
  Frequency of visitors of participant at Baseline
Mini-mental state examination of participant | Baseline measurement
  The mini-mental state examination is a 30-point questionnaire that is used to measure cognitive impairment.
Diagnosis of dementia of participant | Baseline measurement
  Assessment of whether the participant has been determined to have dementia.
Diagnosis of Parkinson's disease of participant | Baseline measurement
  Assessment of whether the participant has been determined to have Parkinson's disease.
Diagnosis of cancer of participant | Baseline measurement
  Assessment of whether the participant has been determined to have cancer.
Diagnosis of Chronic obstructive pulmonary disease of participant | Baseline measurement
  Assessment of whether the participant has been determined to have Chronic obstructive pulmonary disease.
Diagnosis of cardiovascular diseases of participant | Baseline measurement
  Assessment of whether the participant has been determined to have cardiovascular diseases.
Diagnosis of cerebral vascular accident of participant | Baseline measurement
  Assessment of whether the participant has been determined to have cerebral vascular accident.
Diagnosis of diabetes of participant | Baseline measurement
  Assessment of whether the participant has been determined to have diabetes.
Diagnosis of depression of participant | Baseline measurement
  Assessment of whether the participant has been determined to have depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Curando vzw, Wingene, West-Vlaanderen, Belgium